CLINICAL TRIAL: NCT01809327
Title: A Randomized, Double-Blind, 5-Arm, Parallel-Group, 26-Week, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin in Combination With Metformin as Initial Combination Therapy in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control With Diet and Exercise
Brief Title: A Study to Evaluate the Effectiveness, Safety, and Tolerability of Canagliflozin in Combination With Metformin in the Treatment of Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100034; 28431754DIA3011 (Other: Janssen Research & Development, LLC); 2011-000400-17 (EudraCT Number)
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Canagliflozin (JNJ-28431754); Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (5):
- Canagliflozin 100 mg (Experimental): Participants will receive one 100 mg canagliflozin capsule before the morning meal and one matching placebo capsule with the evening meal plus placebo tablets with the evening meal (to match the metformin XR tablets administered in other treatment arms) for 26 weeks.
  Interventions: Drug: Canagliflozin 100 mg
- Canagliflozin 300 mg (Experimental): Participants will receive one 300 mg canagliflozin capsule before the morning meal and one matching placebo capsule with the evening meal plus placebo tablets with the evening meal (to match the metformin XR tablets administered in other treatment arms) for 26 weeks.
  Interventions: Drug: Canagliflozin 300 mg
- Metformin XR (Experimental): Participants will receive metformin XR tablets (in doses titrated over 9 weeks) once daily with the evening meal, plus one placebo capsule before the morning meal and one placebo capsule with the evening meal (to match the canagliflozin capsules administered in other treatment arms) for 26 weeks.
  Interventions: Drug: Metformin XR
- Canagliflozin 100 mg + Metformin XR (Experimental): Participants will receive one 100 mg canagliflozin capsule with the evening meal and one matching placebo capsule before the morning meal plus metformin XR tablets (in doses titrated over 9 weeks) once daily with the evening meal for 26 weeks.
  Interventions: Drug: Canagliflozin 100 mg; Drug: Metformin XR
- Canagliflozin 300 mg + Metformin XR (Experimental): Participants will receive one 300 mg canagliflozin capsule with the evening meal and one matching placebo capsule before the morning meal plus metformin XR tablets (in doses titrated over 9 weeks) once daily with the evening meal for 26 weeks.
  Interventions: Drug: Canagliflozin 300 mg; Drug: Metformin XR

INTERVENTIONS:
Drug: Canagliflozin 100 mg — One 100 mg capsule taken orally (by mouth) once daily either before the morning meal (for the Canagliflozin 100 mg arm) or with the evening meal (for the Canagliflozin 100 mg + Metformin XR arm).
  Arms: Canagliflozin 100 mg; Canagliflozin 100 mg + Metformin XR
Drug: Canagliflozin 300 mg — One 300 mg capsule taken orally (by mouth) once daily either before the morning meal (for the Canagliflozin 300 mg arm) or with the evening meal (for the Canagliflozin 300 mg + Metformin XR arm).
  Arms: Canagliflozin 300 mg; Canagliflozin 300 mg + Metformin XR
Drug: Metformin XR — One 500 mg tablet (Day 1 up to week 1); two 500 mg tablets (Week 1 up to Week 3); three 500 mg tablets (Week 3 to Week 6); four 500 mg tablets (Week 6 to Week 9). Tablets will be administered with the evening meal.
  Arms: Canagliflozin 100 mg + Metformin XR; Canagliflozin 300 mg + Metformin XR; Metformin XR

SUMMARY:
The purpose of this study is to assess the effectiveness of the co-administration of canagliflozin and metformin extended release (XR) compared with canagliflozin alone, and metformin XR alone in patients with type 2 diabetes mellitus with inadequate control despite treatment with diet and exercise. The safety and tolerability of canagliflozin will also be assessed.

DETAILED DESCRIPTION:
This study will be a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), active-controlled (one of the treatments is an established effective treatment for type 2 diabetes mellitus), parallel-group (each group of participants will be treated at the same time), 5-arm (groups), multicenter study. Approximately 1,200 participants will be randomly assigned to the 5 treatment arms in a 1:1:1:1:1 ratio for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have type 2 diabetes mellitus with inadequate glycemic control on diet and exercise
* Not on antihyperglycemic agent therapy (at least 12 weeks before screening) and have a screening visit fingerstick glycated hemoglobin (HbA1c) of more than or equal to 7 percent and less than or equal to 12.5 percent
* Have a screening visit HbA1c of more than or equal to 7.5 percent and less than or equal to 12 percent as determined by the central laboratory
* Must have a fasting plasma glucose of less than or equal to 300 mg/dL (16.7 mmol/L) prior to randomization
* Must have a fasting fingerstick glucose of greater than 120 mg/dL (6.7 mmol/L) performed at home or at the study center prior to randomization

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Fasting C-peptide less than 0.70 ng/mL (0.23 nmol/L) in participants for whom the investigator cannot reasonably exclude T1DM based upon clinical evaluation
* Repeated (2 or more over a 1 week period) fasting self-monitored blood glucose measurements more than 300 mg/dL (16.7 mmol/L) prior to randomization, despite reinforcement of diet and exercise counseling
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria
* Has history of, or currently active, illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2013-06-04 (Actual); Primary Completion 2014-12-02 (Actual); Study Completion 2014-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (129):
- United States (52):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Encinitas, California
  - Newport Beach, California
  - Northridge, California
  - Norwalk, California
  - Rancho Cucamonga, California
  - Walnut Creek, California
  - Denver, Colorado
  - Northglenn, Colorado
  - Hialeah, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Opa-locka, Florida
  - Perry, Georgia
  - Evansville, Indiana
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - Sunset, Louisiana
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Olive Branch, Mississippi
  - Picayune, Mississippi
  - Albuquerque, New Mexico
  - West Seneca, New York
  - Hickory, North Carolina
  - Mooresville, North Carolina
  - Franklin, Ohio
  - Mason, Ohio
  - Perrysburg, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Yukon, Oklahoma
  - Tualatin, Oregon
  - Fleetwood, Pennsylvania
  - Norristown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Austin, Texas
  - Bellaire, Texas
  - Dallas, Texas
  - Houston, Texas
  - Pearland, Texas
  - Plano, Texas
  - Bountiful, Utah
  - Salt Lake City, Utah
  - Danville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
- Argentina (7):
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Córdoba
  - Mar del Plata
  - Morón
  - Rosario
  - Zárate
- Brazil (2):
  - Passo Fundo
  - São Paulo
- Czechia (4):
  - Kroměříž
  - Pardubice
  - Prague
  - Uničov
- Hungary (5):
  - Balatonfüred
  - Budapest
  - Eger
  - Szikszó
  - Zalaegerszeg
- Mexico (7):
  - Celaya
  - Durango
  - Guadalajara
  - México
  - Monterrey
  - Pachuca
  - Tampico
- Puerto Rico (4):
  - Carolina
  - Ponce
  - San Juan
  - Trujillo Alto
- Romania (5):
  - Bacau
  - Brasov
  - Bucharest
  - Oradea
  - Tg Mures
- Russia (15):
  - Arkhangelsk
  - Barnaul
  - Chelyabinsk
  - Kemerovo
  - Moscow
  - Penza
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Saratov
  - Smolensk
  - Syktyvkar
  - Tomsk
  - Tyumen
  - Voronezh
- Slovakia (7):
  - Banská Bystrica
  - Bratislava
  - Malacky
  - Prešov
  - Rimavská Sobota
  - Šahy
  - Trebišov
- South Africa (6):
  - Cape Town
  - Durban
  - Halfway
  - Johannesburg
  - Soweto, Johannesburg
  - Worcester
- South Korea (3):
  - Goyang-si
  - Seoul
  - Suwon
- Ukraine (12):
  - Cherkasy
  - Dnipro
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Sumy
  - Zaporizhzhya

REFERENCES:
- [Derived] Rosenstock J, Chuck L, Gonzalez-Ortiz M, Merton K, Craig J, Capuano G, Qiu R. Initial Combination Therapy With Canagliflozin Plus Metformin Versus Each Component as Monotherapy for Drug-Naive Type 2 Diabetes. Diabetes Care. 2016 Mar;39(3):353-62. doi: 10.2337/dc15-1736. Epub 2016 Jan 19. PMID 26786577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 16 May 2013 and 01 December 2014 and recruited participants from 158 study centers in 12 countries worldwide.
Pre-assignment Details: A total of 1,186 participants were randomly allocated to the 5 treatment arms. All participants received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set.
Groups:
- Metformin XR: Participants received metformin extended release (XR) tablets (in doses titrated over 9 weeks) once daily with the evening meal, plus one placebo capsule before the morning meal and one placebo capsule with the evening meal (to match the canagliflozin capsules administered in other treatment arms) for 26 weeks.
- Canagliflozin 100 Milligram (mg): Participants received one 100 milligram (mg) canagliflozin capsule before the morning meal and one matching placebo capsule with the evening meal plus placebo tablets with the evening meal (to match the metformin XR tablets administered in other treatment arms) for 26 weeks.
- Canagliflozin 300 mg: Participants received one 300 mg canagliflozin capsule before the morning meal and one matching placebo capsule with the evening meal plus placebo tablets with the evening meal (to match the metformin XR tablets administered in other treatment arms) for 26 weeks.
- Canagliflozin 100 mg + Metformin XR: Participants received one 100 mg canagliflozin capsule with the evening meal and one matching placebo capsule before the morning meal plus metformin XR tablets (in doses titrated over 9 weeks) once daily with the evening meal for 26 weeks.
- Canagliflozin 300 mg + Metformin XR: Participants received one 300 mg canagliflozin capsule with the evening meal and one matching placebo capsule before the morning meal plus metformin XR tablets (in doses titrated over 9 weeks) once daily with the evening meal for 26 weeks.
Period: Overall Study
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Started | 237 | 237 | 238 | 237 | 237
Completed | 205 | 211 | 216 | 225 | 212
Not Completed | 32 | 26 | 22 | 12 | 25
Not completed — Lost to Follow-up | 5 | 2 | 4 | 2 | 3
Not completed — Withdrawal by Subject | 6 | 4 | 4 | 2 | 5
Not completed — Adverse Event | 4 | 3 | 7 | 4 | 8
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Other | 14 | 15 | 7 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR | Total
Number analyzed (Participants) | 237 | 237 | 238 | 237 | 237 | 1186
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.75) | 54.0 (10.70) | 55.8 (9.56) | 54.2 (9.58) | 55.4 (9.84) | 54.9 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 132 | 113 | 129 | 122 | 617
  Male | 116 | 105 | 125 | 108 | 115 | 569
Region of Enrollment [Number; unit: participants]
  Argentina | 12 | 19 | 21 | 17 | 20 | 89
  Brazil | 1 | 2 | 1 | 0 | 0 | 4
  Czech Republic | 8 | 6 | 6 | 6 | 8 | 34
  Hungary | 2 | 5 | 8 | 9 | 4 | 28
  Mexico | 33 | 31 | 19 | 38 | 38 | 159
  Romania | 24 | 16 | 21 | 27 | 14 | 102
  Russian Federation | 38 | 38 | 45 | 44 | 37 | 202
  Slovakia | 17 | 12 | 22 | 9 | 9 | 69
  South Africa | 5 | 5 | 4 | 5 | 3 | 22
  South Korea | 4 | 2 | 2 | 1 | 3 | 12
  Ukraine | 50 | 56 | 42 | 40 | 54 | 242
  United States | 43 | 45 | 47 | 41 | 47 | 223

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin (HbA1c) From Baseline at Week 26
Description: The change in the value of glycated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) from baseline at Week 26 was compared between the different treatment groups.
Time Frame: Day 1 (Baseline) and Week 26
Population: This analysis was conducted using the modified intent-to-treat analysis set, which included all participants who were randomly assigned to a treatment group and received at least 1 dose of study drug. Here "N" (Number of Participants Analyzed) signifies number of Participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Number analyzed (Participants) | 230 | 230 | 234 | 235 | 236
percentage of hemoglobin | -1.30 (0.071) | -1.37 (0.071) | -1.42 (0.070) | -1.77 (0.069) | -1.78 (0.070)
Statistical Analysis 1: Comparison: Metformin XR vs Canagliflozin 100 mg + Metformin XR; Test type: Superiority or Other; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -0.46, 95% CI 2-sided [-0.657 to -0.269], Standard Error of Mean 0.099
Statistical Analysis 2: Comparison: Metformin XR vs Canagliflozin 300 mg + Metformin XR; Test type: Superiority or Other; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -0.48, 95% CI 2-sided [-0.670 to -0.280], Standard Error of Mean 0.099
Statistical Analysis 3: Comparison: Canagliflozin 100 Milligram (mg) vs Canagliflozin 100 mg + Metformin XR; Test type: Superiority or Other; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -0.40, 95% CI 2-sided [-0.594 to -0.207], Standard Error of Mean 0.099
Statistical Analysis 4: Comparison: Canagliflozin 300 mg vs Canagliflozin 300 mg + Metformin XR; Test type: Superiority or Other; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -0.36, 95% CI 2-sided [-0.557 to -0.169], Standard Error of Mean 0.099
Statistical Analysis 5: Comparison: Metformin XR vs Canagliflozin 100 Milligram (mg); Test type: Non-Inferiority or Equivalence — P value corresponds to a comparison that canagliflozin is noninferior to Metformin XR by a margin of 0.35%; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -0.06, 95% CI 2-sided [-0.258 to 0.133], Standard Error of Mean 0.100
Statistical Analysis 6: Comparison: Metformin XR vs Canagliflozin 300 mg; Test type: Non-Inferiority or Equivalence — P value corresponds to a comparison that canagliflozin is noninferior to Metformin XR by a margin of 0.35%; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -0.11, 95% CI 2-sided [-0.307 to 0.082], Standard Error of Mean 0.099

2. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 26
Description: The percentage change in body weight from baseline to Week 26 was compared between the different treatment groups.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Number analyzed (Participants) | 237 | 236 | 236 | 237 | 236
percent change | -2.1 (0.3) | -3.0 (0.3) | -3.9 (0.3) | -3.5 (0.3) | -4.2 (0.3)
Statistical Analysis 1: Comparison: Metformin XR vs Canagliflozin 100 Milligram (mg); Test type: Superiority or Other; p = 0.016, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -0.9, 95% CI 2-sided [-1.6 to -0.2], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Metformin XR vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.002, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -1.8, 95% CI 2-sided [-2.6 to -1.1], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Metformin XR vs Canagliflozin 100 mg + Metformin XR; Test type: Superiority or Other; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -1.4, 95% CI 2-sided [-2.1 to -0.6], Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: Metformin XR vs Canagliflozin 300 mg + Metformin XR; Test type: Superiority or Other; p = 0.001, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -2.1, 95% CI 2-sided [-2.9 to -1.4], Standard Error of Mean 0.4

3. Secondary Outcome: Percentage of Participants With Glycated Hemoglobin (HbAIc) Less Than 7 Percent at Week 26
Description: The percentage of participants achieved HbAIc less than 7 percent at Week 26 was compared between the different treatment groups.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Number analyzed (Participants) | 207 | 206 | 215 | 224 | 213
percentage of participants | 43.0 | 38.8 | 42.8 | 49.6 | 56.8
Statistical Analysis 1: Comparison: Metformin XR vs Canagliflozin 100 mg + Metformin XR; Test type: Superiority or Other; p = 0.027, Generalized Linear Mixed Model; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.06 to 2.37]
Statistical Analysis 2: Comparison: Metformin XR vs Canagliflozin 300 mg + Metformin XR; Test type: Superiority or Other; p = 0.016, Generalized Linear Mixed Model; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.46 to 3.33]

4. Secondary Outcome: Change in Systolic Blood Pressure From Baseline at Week 26
Description: The change in systolic blood pressure from baseline at Week 26 was compared between the different treatment groups.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mm Hg)
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Number analyzed (Participants) | 237 | 236 | 236 | 237 | 236
millimeter of mercury (mm Hg) | -0.33 (0.633) | -2.24 (0.627) | -2.36 (0.622) | -2.24 (0.613) | -1.65 (0.624)
Statistical Analysis 1: Comparison: Metformin XR vs Canagliflozin 100 mg + Metformin XR; Test type: Superiority or Other; p = 0.060, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -1.91, 95% CI 2-sided [-3.641 to -0.182], Standard Error of Mean 0.882
Statistical Analysis 2: Comparison: Metformin XR vs Canagliflozin 300 mg + Metformin XR; Test type: Superiority or Other; p = 0.147, Mixed Model for Repeated Measures (MMRM); Least-Squares Mean Difference = -1.31, 95% CI 2-sided [-3.058 to 0.431], Standard Error of Mean 0.889

5. Secondary Outcome: Percent Change in Fasting High-Density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26
Description: The percentage change in Fasting High-Density Lipoprotein Cholesterol (HDL-C) from baseline to Week 26 was compared between the different treatment groups.
Time Frame: Day 1 (Baseline) and Week 26
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Here "N" (Number of Participants Analyzed) signifies number of Participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Number analyzed (Participants) | 222 | 225 | 228 | 227 | 225
percent change | 10.2 (1.5) | 17.6 (1.5) | 16.6 (1.5) | 15.5 (1.5) | 14.5 (1.5)
Statistical Analysis 1: Comparison: Metformin XR vs Canagliflozin 100 mg + Metformin XR; Test type: Superiority or Other; p = 0.147, ANCOVA; Least-Squares Mean Difference = 5.3, 95% CI 2-sided [1.2 to 9.5], Standard Error of Mean 2.1
Statistical Analysis 2: Comparison: Metformin XR vs Canagliflozin 300 mg + Metformin XR; Test type: Superiority or Other; p = 0.147, ANCOVA; Least-Squares Mean Difference = 4.3, 95% CI 2-sided [0.2 to 8.5], Standard Error of Mean 2.1

6. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 26
Description: The percentage change in triglycerides from baseline to Week 26 was compared between the different treatment groups.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Number analyzed (Participants) | 223 | 225 | 229 | 229 | 225
percent change | 13.6 (51.8) | 1.7 (50.5) | 2.8 (60.3) | 13.0 (81.9) | 21.2 (71.1)
Statistical Analysis 1: Comparison: Metformin XR vs Canagliflozin 100 mg + Metformin XR; Test type: Superiority or Other; p = 0.608, Wilcoxon (Mann-Whitney); Hodges-Lehman Estimate = -3.7, 95% CI 2-sided [-11.1 to 3.4]
Statistical Analysis 2: Comparison: Metformin XR vs Canagliflozin 300 mg + Metformin XR; Test type: Superiority or Other; p = 0.806, Wilcoxon (Mann-Whitney); Hodges-Lehman Estimate = 1.3, 95% CI 2-sided [-7.3 to 10.0]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study drug and up to 30 days after last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Up to 30 weeks of last study drug administration
Population: Safety Analysis Set included all randomized participants who received at least 1 dose of double-blind study drug.
Measure: Number; unit: participants
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Number analyzed (Participants) | 237 | 237 | 238 | 237 | 237
participants | 89 | 88 | 95 | 99 | 105

ADVERSE EVENTS:
Time Frame: Up to 30 weeks of last study drug administration
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Event" table are based on atleast 2 percent of participants experiencing the adverse event in any treatment arm.
Arm/Group | Metformin XR | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Canagliflozin 100 mg + Metformin XR | Canagliflozin 300 mg + Metformin XR
Serious Adverse Events (participants affected / at risk) | 7/237 | 4/237 | 7/238 | 7/237 | 4/237
Other Adverse Events (participants affected / at risk) | 37/237 | 38/237 | 38/238 | 42/237 | 43/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin XR (N=237) | Canagliflozin 100 Milligram (mg) (N=237) | Canagliflozin 300 mg (N=238) | Canagliflozin 100 mg + Metformin XR (N=237) | Canagliflozin 300 mg + Metformin XR (N=237)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Epiploic Appendagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cardiac Death (General disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ophthalmic Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Extradural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Medullary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Arterial Occlusive Disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin XR (N=237) | Canagliflozin 100 Milligram (mg) (N=237) | Canagliflozin 300 mg (N=238) | Canagliflozin 100 mg + Metformin XR (N=237) | Canagliflozin 300 mg + Metformin XR (N=237)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 4 | 10 | 10
Nausea (Gastrointestinal disorders) | 6 | 1 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 2 | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 1 | 1 | 5
Influenza (Infections and infestations) | 5 | 6 | 5 | 8 | 7
Nasopharyngitis (Infections and infestations) | 3 | 9 | 9 | 6 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 2 | 6 | 3 | 4
Urinary Tract Infection (Infections and infestations) | 3 | 3 | 4 | 2 | 7
Glomerular Filtration Rate Decreased (Investigations) | 0 | 6 | 3 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 5 | 1 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5 | 6 | 5
Headache (Nervous system disorders) | 8 | 4 | 4 | 9 | 7
Hypertension (Vascular disorders) | 1 | 2 | 2 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.